CLINICAL TRIAL: NCT05657613
Title: Drug-Drug Interaction Study of Multiple Doses of Pacritinib and CYP450 And, Transporter Substrates, and CYP450 3A4 Inducers and Inhibitors
Brief Title: Drug-Drug Interaction Study of Pacritinib and CYP450,Transporter Substrates, and CYP450 3A4 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAC109
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Drug Interactions
Keywords: Pacritinib; Cytochrome P450 and Transporters
MeSH Terms: interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Intervention Model Description: An open-label, fixed-sequence, 2-part drug-drug interaction study of pacritinib in healthy adult males
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- CYP450 Cocktail and Transporter Substrates with Pacritinib (Experimental): This is the first part of the study which is an open-label, single-center, 1-way DDI study designed to assess the effect of pacritinib 200 mg BID at steady state on the systemic exposure of a cocktail of cytochrome P450 (caffeine, midazolam, and omeprazole) and transporter substrates (digoxin, rosuvastatin, and metformin) in 18 healthy male subjects.
  Interventions: Drug: CYP450 Cocktail and Transporter Substrates with Pacritinib
- CYP450 3A4 inducer (Bosentan) with Pacritinib (Experimental): The second part of the study comprises of 2 arms. This is the first arm Days 1 through 14: An oral dose of pacritinib 200 mg (2 × 100 mg capsules) BID (approximately 12 hours apart) Days 8 through 14: An oral dose of bosentan 125 mg BID (approximately 12 hours apart) All the doses will be administered with approximately 240 mL of water.
  Interventions: Drug: Part 2 -Group A Bosentan 125 mg (CYP450 3A4 inducer) with Pacritinib
- CYP450 3A4 inhibitor (Fluconazole) with Pacritinib (Experimental): This is the second arm of Part 2 of the study:
  Days 1 through 14: An oral dose of pacritinib 200 mg (2 × 100 mg capsules) BID (approximately 12 hours apart) Days 8 through 14: An oral dose of fluconazole 200 mg QD
  Interventions: Drug: Part 2 Group B - Fluconazole (CYP450 3A4 inhibitor) with Pacritinib

INTERVENTIONS:
Drug: CYP450 Cocktail and Transporter Substrates with Pacritinib — Day 1: Single oral dose of a cocktail of cytochrome P450 substrates (caffeine 100 mg, midazolam 2 mg, omeprazole 20 mg and metformin (transporter)
  Day 3: Single oral dose of transporter substrates (digoxin 0.25 mg, rosuvastatin 5 mg)
  Days 8-22: Oral doses of pacritinib 200 mg BID approximately 12 hours apart
  Day 17: Single oral dose of transporter substrates (digoxin 0.25 mg and rosuvastatin 5 mg) will be coadministered with the AM dose of pacritinib 200 mg.
  Day 21: Single oral dose of a cocktail of cytochrome P450 substrates (caffeine 100 mg, midazolam 2 mg, and omeprazole 20 mg) along with transporter substrate (metformin 500 mg) will be coadministered with the AM dose of pacritinib 200 mg.
  Other Names: Vonjo
  Arms: CYP450 Cocktail and Transporter Substrates with Pacritinib
Drug: Part 2 -Group A Bosentan 125 mg (CYP450 3A4 inducer) with Pacritinib — Days 1-7: Oral doses of pacritinib 200 mg BID
  Days 8-14: Oral doses of pacritinib 200 mg BID, coadministered with an oral dose of bosentan 125 mg BID
  Other Names: Vonjo
  Arms: CYP450 3A4 inducer (Bosentan) with Pacritinib
Drug: Part 2 Group B - Fluconazole (CYP450 3A4 inhibitor) with Pacritinib — Days 1-7: Oral doses of pacritinib 200 mg BID
  Days 8-14: Oral doses of pacritinib 200 mg BID, coadministered with an oral dose of fluconazole 200 mg QD.
  Other Names: Vonjo
  Arms: CYP450 3A4 inhibitor (Fluconazole) with Pacritinib

SUMMARY:
This is a Phase 1, open-label, fixed-sequence, 2-part DDI study. Subjects will participate in only 1 study part.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, fixed-sequence, 2-part DDI study. Part 1 will evaluate the effect of 14 days of pacritinib 200 mg BID at steady state on the systemic exposure of a cocktail of single doses of cytochrome P450 (caffeine, midazolam, omeprazole) and transporter substrates (digoxin, rosuvastatin, metformin) in 18 healthy male subjects who will participate in 2 treatment periods sequentially separated by a washout period. Part 2 will evaluate the effect of a CYP450 3A4 inducer (bosentan BID) for 7 days and the effect of a CYP450 3A4 inhibitor (fluconazole QD) for 7 days, on the PK of multiple doses of pacritinib 200 mg BID in 36 healthy male subjects. Safety and tolerability will be assessed by AEs, clinical laboratory tests, vital signs, ECGs, and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male 18 to 55 years of age, inclusive, at screening.
* The subject has a BMI of 18.0 to 32.0 kg/m2, inclusive, at screening.
* The subject has a normal renal function ≥60 mL/min eGFR.
* The subject is considered by the investigator to be in good general health as determined by medical history review, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings at screening and check-in.
* The male subjects will be sterile, or completely abstain from sexual intercourse, or agree to use, from check-in (Day -1) until 90 days following EOS/ET, one of the following approved methods of contraception: male condom with spermicide or a sterile sexual partner; or use by female sexual partner of an IUD with spermicide, a female condom with spermicide, a contraceptive sponge with spermicide, an intravaginal system, a diaphragm with spermicide, a cervical cap with spermicide, or oral, implantable, transdermal, or injectable contraceptives. The subject will refrain from sperm donation from check-in (Day -1) until 90 days following study completion (Day 31 for Part 1 and Day 24 for Part 2).
* The subject must have adequate venous access for blood draws.
* The subject agrees to comply with all protocol requirements.
* The subject is able to provide written informed consent.

Additional Inclusion Criteria for Part 1:

• The subject has a documented result of genotype testing for CYP2C19 *1/*1 suggesting normal metabolizers.

Exclusion Criteria:

* The subject has a history of any clinically significant conditions including the following:
* Asthma treated with oral systemic steroids within the past 6 months
* Diabetes mellitus (types 1 or 2), with the exception of gestational diabetes
* Thyroidectomy or thyroid disease that required medication within the past 12 months
* Serious angioedema episodes within the previous 3 years or requiring medication in the previous 2 years
* Head trauma resulting in a diagnosis of traumatic brain injury other than concussion
* Known clinically relevant history or presence of significant respiratory (eg, interstitial lung disease), GI (eg, GI ulceration, peptic ulceration, GI bleeding, gastroesophageal reflux, or other GI disease affecting gastroesophageal junction), renal, hepatic (eg, known hepatic or biliary abnormalities), hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, metabolic (eg, diabetes) and dermatological or connective tissue disease.
* The subject has a value >1.5 × ULN for any of the following: prothrombin time, partial thromboplastin time, and international normalized ratio.
* The subject has a seated systolic blood pressure >160 mm Hg or ≤90 mm Hg and a diastolic blood pressure of >100 mm Hg or ≤50 mm Hg, inclusive, at screening and check-in unless deemed not clinically significant by the investigator, as approved by the sponsor.
* The subject has a seated pulse rate of <50 bpm or >100 bpm and/or an oral body temperature <35.0°C or >37.5°C when vital signs are measured at screening and check-in.
* The subject has a clinically significant illness, including viral syndromes, within 3 weeks of dosing.
* The subject has a known clinically significant chronic viral infection (eg, human T-cell lymphotropic virus I or II).
* The subject has a history or clinical manifestation of clinically significant cardiovascular, pulmonary, hepatic (eg, hepatitis), renal, hematologic, gastrointestinal (eg, celiac disease, peptic ulcer, gastroesophageal reflux, inflammatory bowel disease), metabolic, allergic, dermatological, neurological, or psychiatric disorder (as determined by the investigator; appendectomy and cholecystectomy [within 3 to 6 months] are not considered to be clinically significant procedures).
* The subject has a history of cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or risk factors for torsades de pointes (eg, heart f failure, hypokalemia).
* The subject has evidence or a history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of the first dose of study drug), hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease. Exceptions to this criterion (eg, stable, mild joint disease unassociated with collagen vascular disease) may be made following discussions with the medical monitor.
* The subject has evidence of neutropenia or any other blood dyscrasia determined to be clinically significant by the investigator.
* The subject has history of a gastrointestinal bleeding.
* The subject has a history of a bleeding disorder diagnosed by a doctor (eg, coagulation factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with blood draws.
* The subject has receipt of blood products within 2 months prior to check-in (Day -1).
* The subject has donated blood or blood products >450 mL within 30 days before the first dose of study drug.
* The subject is a smoker or has used nicotine or nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) within 6 months before the first dose of study drug.
* The subject has a positive test result for drugs of abuse, alcohol, or cotinine (indicating active current smoking) at screening, check-in, or throughout the study.
* The subject has a history or presence of an abnormal ECG, which, in the investigator's opinion, is clinically significant; QTcF >450 msec, or factors that increase the risk for QTc interval prolongation (eg, heart failure, hypokalemia [defined as serum potassium <3.0 mEq/L that is persistent and refractory to correction], or a history of long QT interval syndrome).
* The subject has a history of relevant drug and/or food allergies (ie, allergy to digoxin, caffeine, midazolam, omeprazole, rosuvastatin, metformin, bosentan, and fluconazole or excipients) or a previous allergic reaction to phenytoin or carbamazepine (applicable for Group B subjects).
* The subject has a history of lymphoma, leukemia or other types of malignancy.
* The subject has a current or recent (<30 days before screening) history of clinically significant bacterial, fungal, or mycobacterial infection.
* The subject has a current or recent (<30 days before screening) history of vitamin B12 deficiency.
* The subject is unable to tolerate oral medication.
* The subject has any major surgery within 4 weeks of study drug administration.
* The subject has a family history of sudden cardiac death not clearly due to acute myocardial infarction.
* The subject has any screening or baseline laboratories outside the normal range and deemed clinically significant.
* The subject has used any prescription or over-the-counter medications, including herbal or nutritional supplements, within 14 days of check-in.
* The subject has any condition possibly affecting drug absorption (eg, previous surgery on the gastrointestinal tract, including removal of parts of the stomach, bowel, liver, gallbladder, or pancreas, with the exception of appendectomy).
* The subject has used any of the prohibited medications (targeted CYP inducers or inhibitors) from within 15 days (or 5 half-lives, whichever is longer) before the first dose of study drug.
* The subject has consumed grapefruit or grapefruit juice, Seville orange or Seville orange- containing products (eg, marmalade), or caffeine- or xanthine-containing products or other CYP3A4 inhibitors, inducers, or transporter substrates within 48 hours before the first dose of study drug and throughout the study.
* The subject has consumed pomegranate or pomegranate juice, pomelo fruits or pomelo juice, or alcohol within 72 hours before check-in on Day -1.
* The subject has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies at screening.
* The subject is involved in strenuous activity or contact sports within 24 hours before the first dose of study drug and throughout the study.
* The subject has received treatment in another clinical study of an investigational drug (or medical device) or investigational vaccine within 30 days or 5 half-lives (whichever is longer) prior to check-in.
* The subject has previously received pacritinib.
* The subject is not suitable for entry into the study in the opinion of the investigator.
* Use of any other prescription medications and/or products within 14 days prior to check-in (Day -1) and during the entire study, unless deemed acceptable by the investigator in consultation with the sponsor. In addition, use of any over-the-counter, non-prescription preparations (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) from 7 days prior to check-in (Day -1) and during the entire study, unless deemed acceptable by the investigator.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Change in area under curve (AUC) of individual substrates between cocktail alone and cocktail combined with pacritinib administration | Through study completion, a maximum of 14 days for pacritinib
  Change in the systemic exposure of digoxin, midazolam omeprazole, rosuvastatin, caffeine and metformin when co-adminstered with pacritinib
Change in maximum plasma concentration (Cmax) of individual substrates between cocktail alone and cocktail combined with pacritinib administration | Through study completion, a maximum of 14 days for pacritinib
  To assess the effect of pacritinib on the systemic exposure of digoxin, midazolam, omeprazole, rosuvastatin, caffeine, and metformin
Change in area under curve (AUC) of pacritinib alone and pacritinib + bosentan administration | Through completion, a maximum of 14 days for pacritinib
  To assess the effect of bosentan (CYP450 3A4 inducer) on the systemic exposure of multiple doses of pacritinib
Change in Cmax of pacritinib alone and pacritinib + bosentan administration | Through study completion, a maximum of 14 days for pacritinib
  To assess the effect of bosentan (CYP450 3A4 inducer) on the peak exposure of multiple doses of pacritinib
Change in AUC of pacritinib alone and pacritinib + fluconazole administration | Through study completion, a maximum of 14 days for pacritinib
  To assess the effect of fluconazole (CYP450 3A4 inhibitor) on the systemic exposure of multiple doses of pacritinib
Change in Cmax of pacritinib alone and pacritinib + fluconazole administration | Through study completion, a maximum of 14 days for pacritinib
  To assess the effect of fluconazole (CYP450 3A4 inhibitor) on the systemic peak exposure of multiple doses of pacritinib

SECONDARY OUTCOMES:
Number and severity of adverse events with cocktail substrates in the presence of pacritinib | Up to 31 days
  Any adverse event will be monitored and recorded (including an abnormal clinical laboratory results, an abnormal electrocardiogram), symptom or diseases temporarily associated with the use of a study drug, whether considered related to study drug or not. To assess safety and tolerability of multiple doses of pacritinib coadministered with digoxin, caffeine, midazolam, omeprazole, rosuvastatin, and metformin in healthy male subjects.
Number and severity of adverse events with pacritinib in the presence of CYP450 3A4 inducer | Up to 31 days
  Any adverse event will be monitored and recorded (including an abnormal clinical laboratory results, an abnormal electrocardiogram), symptom or diseases temporarily associated with the use of a study drug, whether considered related to study drug or not. To assess safety and tolerability of multiple doses of pacritinib coadministered with bosentan in healthy male subjects.
Number and severity of adverse events with pacritinib in the presence of CYP450 3A4 inhibitor | Up to 31days
  Any adverse event will be monitored and recorded (including an abnormal clinical laboratory result, an abnormal electrocardiogram), symptom or diseases temporarily associated with the use of a study drug, whether considered related to study drug or not. To assess safety and tolerability of multiple doses of pacritinib coadministered with fluconazole in healthy male subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Buckley, Study Director — CTI BioPharma
Locations (1):
- Site 1, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No